CLINICAL TRIAL: NCT00629421
Title: Early Screening of Hepatocellular Carcinoma in Cirrhotic Patients: a Prospective Study
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jung-Fa,Tsai, Professor of Medicine, Kaohsiung Medical University Chung-Ho Memorial Hospital
Other Study IDs: KMUH-IRB-960012
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Cirrhosis; Hepatocellular Carcinoma
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Although serum alpha-fetoprotein level and abdominal sonography are the main methods to screening hepatocellular carcinoma (HCC) in cirrhotic patients, the adequate time and methods used are not completely well-defined. This study aims to assess the better timing and methods for prospectively screening HCC in patients with cirrhosis

DETAILED DESCRIPTION:
Well-diagnosed consecutive patients with cirrhosis were enrolled through a designed questionnaire to obtain basic information about gender, age, etiology of cirrhosis, conventional liver function tests, serum AFP level, education level, substance use including smoking, alcohol drinking, betel quid chewing, history of familial HCC, etc. Then the patients was followed by periodic abdominal sonography examination and determination of AFP and liver function. If AFP elevated or liver nodule appears, effort to diagnose HCC will be performed.If HCC was performed, the survival will be followed-up. As anti-viral therapy was found to decrease risk for HCC, patients with those therapy will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Image diagnosis or biochemical diagnosis or presence of portal hypertension

Exclusion Criteria:

* Presence of hepatocellular carcinoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Well-dignosed patients with cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2001-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
development of hepatocellular carcinoma | during observation
  nodule (with or without seum AFP greater than 400 ng/ml) confirmed by biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Fa Tsai, M.D., Ph.D., Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan